CLINICAL TRIAL: NCT01672190
Title: Lessening Incontinence by Learning Yoga
Acronym: LILY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Alison Huang, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-09389
Record Dates: First submitted 2012-08-16; First posted 2012-08-24 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Urinary Incontinence; Stress Urinary Incontinence; Urge Urinary Incontinence; Over Active Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Therapy (Experimental): Women in the Yoga Therapy Group will receive twice weekly yoga classes for 6 weeks.
  Interventions: Other: Yoga Therapy Program
- Control (No Intervention): Women in the Control Group will wait 6 weeks before receiving a gift certificate for yoga classes at an external yoga studio in the San Francisco Bay Area

INTERVENTIONS:
Other: Yoga Therapy Program
  Arms: Yoga Therapy

SUMMARY:
The purpose of this study is to assess the feasibility of recruiting women with urinary incontinence into a randomized controlled trial of a yoga therapy program.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40 years or older who report urinary incontinence for > 3 months prior to screening
* Self-report at least 7 urinary incontinence episodes per week on a screening 7-day voiding diary
* Self-report urgency-predominant, stress-predominant, or mixed-type incontinence on the screening voiding diary
* Willing to refrain from initiating medical treatments that may affect their incontinence or voiding pattern during the study period
* Capable of understanding study procedures and giving informed consent

Exclusion Criteria:

* Participation in a yoga class or other formal or organized yoga instruction in the past year
* Any prior yoga therapy directed specifically at improving urinary incontinence or pelvic floor dysfunction
* Current use of medical therapy or device (i.e. pessary) for incontinence or use within the previous month
* Currently pregnant, gave birth within the past 6 months, or planning pregnancy during the study period
* Current urinary tract infection or a history or 3 or more urinary tract infections in the preceding year
* Report history of neurologic conditions such as stroke, multiple sclerosis, spinal cord injury, or Parkinson's disease, or a lumbosacral spine condition associated with neurological symptoms
* Unable to walk up a flight of stairs or at least 2 blocks on level ground without assistance
* Unable to get up from a supine to a standing position in 10 seconds or less and without assistance
* Severe obesity, defined as body mass index > 35 kg/m2 on screening examination
* Report history of interstitial cystitis, fistula or hole in bladder or rectum, or birth defect leading to urine leakage
* Report any history of prior anti-incontinence or urethral surgery (not including urethral dilation), pelvic cancer, or pelvic irradiation for any reason
* Report use of bladder botox, electrostimulation, bladder training, or pelvic floor exercise training (with certified practitioners) in the past 3 months
* Report other surgery to the pelvis (hysterectomy, oophorectomy, vaginal surgery, bladder surgery, colon surgery) within the past 3 months
* Report symptomatic pelvic organ prolapse
* Report history of vulvodynia, chronic pelvic pain, or pain when practicing pelvic floor exercises
* Report conditions that, in the judgment of the investigators, render potential participants unlikely to follow the protocol, including plans to move, substance abuse, significant psychiatric problems, or dementia
* Participation in another research study that involves investigational drugs or devices that could potentially confound the results of this study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in the number of incontinence episodes over 7 days, with 95% confidence intervals, between baseline and 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States